CLINICAL TRIAL: NCT02938117
Title: Impact of a Training Program on the Body Composition of Overweight and Obese Young Adults : Concentric Versus Eccentric Exercise
Acronym: OPEX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: CHU-0284; 2016-A01185-46 (Other: 2016-A01185-46)
Record Dates: First submitted 2016-10-10; First posted 2016-10-19 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Adults; BMI>35
Keywords: obesity; eccentric exercise; body composition; training program
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- CON : concentric cycling exercise (Experimental): Thirty adults will be randomized into 2 groups: CON or EXC. The patients of ECC group will follow habituation sessions (2weeks) to avoid the secondary muscular effects of high intensity eccentric exercise
  Interventions: Other: cycling exercises
- EXC : eccentric cycling exercise (Experimental): Thirty adults will be randomized into 2 groups: CON or EXC. The patients of ECC group will follow habituation sessions (2weeks) to avoid the secondary muscular effects of high intensity eccentric exercise
  Interventions: Other: cycling exercises

INTERVENTIONS:
Other: cycling exercises

SUMMARY:
Nowadays, eccentric exercise can be realized in a dynamic way with an ergocycle wich permits eccentric (ECC) lower limbs contractions at a defined power output. With this type of ergometer, O2 consumption (VO2) in ECC is three fold lower than in concentric (CON) for the same power output. Consequently, ECC program could be used in chronic disorders with limited capacities, such as obesity.

The investigators hypothesis that an eccentric training program, as it will induce higher mechanical constraints, would improve body composition, especially by reducing fat mass. This effect could be explained by an increased rest energy expenditure and a better improvement in biological parameters (particularly lipid profile and insulin-resistance) after ECC training (versus CON training).

This study aims to compare the modification of fat mass after an ECC program versus a CON program at the same VO2. The secondary goal is to assess the physiological mechanisms involved in the modification of body composition

DETAILED DESCRIPTION:
Thirty adults will be randomized into 2 groups: CON or EXC. The patients of ECC group will follow habituation sessions (2weeks) to avoid the secondary muscular effects of high intensity eccentric exercise. The training program will last 12 weeks for the two groups. Before and after, each subjects will participate to the following measurements: total and segmental body composition (DXA), aerobic capacities (maximal incremental exercise test, VO2max), muscular lower limbs strength (isometric end isokinetic dynamometer), rest energy expenditure (indirect calorimetry), biological parameters (lipid profile, insulin-resistance), physical activity (actimetry), food intakes and quality of life (questionnaires).

ELIGIBILITY:
Inclusion Criteria:

* - Adults
* Obese (BMI>35)
* Inactive (<10 METS/h/week)
* No other chronic disease (cardio pulmonary, osteo articulary or muscular diseases), no surgery during the last 3 months, no contraindication to physical activity

Exclusion Criteria:

* (BMI<35)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-12 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
change in total body fat mass (Dual X ray Absorptiometry) | before and after the 12 weeks training program

SECONDARY OUTCOMES:
aerobic capacities (VO2max) | before and after the 12 weeks training program
isometric muscular lower limbs strength | before and after the 12 weeks training program
isokinetic muscular lower limbs strength | before and after the 12 weeks training program
rest energy expenditure (indirect calorimetry) | before and after the 12 weeks training program
biological parameters (plasma lipid profile) | before and after the 12 weeks training program
biological parameters (insulin-resistance) | before and after the 12 weeks training program
physical activity | before and after the 12 weeks training program
  (questionnaires)
physical activity | before and after the 12 weeks training program
  (actimetry)
food intakes | before and after the 12 weeks training program
  (measurements)
food intakes | before and after the 12 weeks training program
  (questionnaires)
quality of life (questionnaires) | before and after the 12 weeks training program
segmental body composition | before and after the 12 weeks training program
  (segmental fat and fat free mass)

CONTACTS AND LOCATIONS:
Overall Officials: Valérie JULIAN, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France